CLINICAL TRIAL: NCT05114824
Title: Pilot Study of the Acceptability and Feasibility of an 8-week Online Mindfulness-Based Cognitive Therapy Programamong Undergraduate Students: a Randomized Controlled Trial
Brief Title: Acceptability and Feasibility of an 8-week Online Mindfulness-Based Cognitive Therapy Program Among Undergraduate Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Ministerio de Educación, Chile (Unknown)
Responsible Party: Principal Investigator, Jorge Gaete, Principal Investigator, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDI UAN1901-1
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Stress, Psychological; Anxiety Disorders; Depression, Unipolar
Keywords: Mindfulness; Students; MBCT; Mindfulness-Based Cognitive Therapy
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depressive Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): Mindfulness-Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Control Group (No Intervention): Control group

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — The intervention is based on a mixed MBCT program with training in mindfulness strategies for 8 weeks. The adapted MBCT intervention will consist of eight weekly group sessions of 1 hour and 30 minutes, led by a certified instructor, to address the symptoms in the university population. In addition, complemented with the inclusion of audiovisual material, aimed at guiding self-applied daily exercises.
  Other Names: MBCT
  Arms: Mindfulness-Based Cognitive Therapy

SUMMARY:
Mental health problems -particularly depression- are the main cause of morbidity in young people (1), which has a known association with different health and social problems, such as increased alcohol consumption and drug dependence, adolescent pregnancy, school dropouts , criminal behavior, self-harm, and even suicide (2-4). MBCT is an intervention that has been shown to reduce depression, stress and anxiety in the adult and university population; however, its duration and time demands make it difficult to implement. The available evidence of mindfulness interventions in university students is heterogeneous, with various methodological flaws, and is based on self-applied programs such as Mindful Mood Balance (MMB), without the participation of instructors.

The current study aim to explore the acceptability and feasibility of an intervention based on a Mindfulness-based Cognitive Therapy (MBCT) program with training in mindfulness strategies for 8 weeks. The adapted MBCT intervention will consist of eight weekly group sessions of 1 hour and 30 minutes, led by a certified instructor, to address the depressive and anxiety symptoms in the university population. In addition, the intervention will be complemented with the inclusion of audiovisual material, aimed at guiding self-applied daily exercises.

DETAILED DESCRIPTION:
1. Study design This is an experimental type study, with a randomized controlled trial design, with a control group in the waiting list mode. The intervention is an synchronous online mindfulness training, lasting eight weeks for university population.
2. Participants:

   The participants will be undergraduate students from the Universidad de los Andes, studying from 2nd to last year, of different careers.
3. Sample size Although this is a pilot study, with the main focus on determining the acceptability and feasibility of a preventive intervention based on mindfulness, a sample calculation is carried out in order to explore the efficacy of this intervention under controlled conditions such as those proposed in this draft. For this calculation, the intensity of depressive symptoms is considered as the main response variable or primary outcome. We will use an effect size of big nature (Cohen's d = 0.8), similar to that found in other pilot studies that evaluated similar interventions. Considering a statistical power of 0.80 and an alpha of 0.05, and according to a two-tailed hypothesis test, we will need 26 participants per group (52 in total). Considering that we expect a loss of about 20% of the participants, the minimum number to recruit in the proposed study will be 62 (31 per group). The intervention proposed in this study can be applied remotely to a maximum of 20 students, so the students will be separated into 2 subgroups that will do the intervention in parallel, for 8 weeks.
4. Process

   4.1. Recruitment The potential participants will be undergraduate students from the Universidad de los Andes, who meet the inclusion and exclusion criteria previously described. They will learn about the study through invitations that will be made to their institutional email and social networks, by the research team, to carry out the study instruments and having signed an informed consent.

   4.1.1 Enrollment Strategy This research project and the mindfulness intervention will be disseminated after the approval of the Scientific Ethics Committee, during the first weeks of the second semester of 2021. It will be disseminated via personal email with the relevant information of the study, in addition a cycle of informative talks ("Seminars"), whose link will be sent via email. The talks will inform about the duration, requirements, benefits, risks of participating in the study. These talks will be conducted by the mindfulness instructors, having total privacy of what is discussed in them. Once the meeting is over, interested persons will be invited to sign the informed consent, fill out the screening instruments and leave their contact information to participate in the intervention. Through these screening instruments, it will be possible to identify students who meet inclusion and exclusion criteria. Students who meet the inclusion criteria will be contacted and the group they belong will be informed according to the randomization procedure. Those students who have a score of ≥15 points on the PHQ-9 scale will not be able to participate in the intervention, and they will be invited to use the intervention "Take care of your mood "(universal intervention that shows beneficial effects for the prevention of depressive symptoms) available for free at the following link (http://cuidatuanimo.net), where you will find useful information to prevent depressive symptoms. This intervention has been developed by a research team with whom Dr Jorge Gaete collaborates. Additionally, they will also be invited to request help in the Unit of Wellbeing of University Life at Universidad de los Andes. This group of students will be contacted by the research team, a week, and 2 weeks after having answered the screening instrument to find out if they requested an appointment with the University Wellbeing team.

   4.1.2. Informed consent Informed consent will be requested from students. The students of the Universidad de los Andes will be invited to participate in an informative seminar about the study. Once the study, inclusion and exclusion criteria have been explained, the exhibitor will provide interested parties with a description of the screening instruments, their importance and selection process. If they accept to participate, the informed consent will be sent to the emails, which will be signed digitally through Qualtrics (A platform that allows information to be collected online, with high-security standards and that also has the ability to facilitate the digital signature through a cell phone or tablet (using the finger) or through a computer (with a mouse), and also the screening instrument that will evaluate: sociodemographic data, depression, anxiety and stress, mindfulness skills, physical and psychiatric comorbidities, prior consultations to mental health services, medications, alcohol and drug use, previous practice of mindfulness, quality of life. These data will be used for the study eligibility analysis. Those who meet the inclusion criteria will be enrolled in the study and they will be randomly distributed in the intervention group and the control group.

   Informed consent will cover both general screening and baseline measurements and follow-up during and after the intervention.

   4.2. Evaluation procedure Measurement of baseline status: The week prior to the start of the intervention, self-report questionnaires (PHQ-9, GAD-7, ASSIST, PROMIS Global Health v1.2, FFMQ, SF-36 v.2), sociodemographic characterization, among others, will be used. As already stated in the previous section, the PHQ-9 will be one of the elements to determine compliance with the inclusion and exclusion criteria.

   4.3. Randomization: All participants who meet the inclusion and exclusion criteria, after granting informed consent, will be randomized to 2 groups, distributing them between the control group or the intervention group. The randomization will be carried out through the "random" formula of an Excel spreadsheet, which allows this random distribution to be carried out. Each group will have about at least 26 participants.

   4.4. Blind condition: By the nature of the intervention, the participants are not blind to the group to which they belong. The evaluations will be carried out through the self-report of questionnaires sent in electronic format and their evaluation will be automatic, without human action. In data analysis, the statistician will be blind to the intervention group of participants.
5. Study duration The entire study, from its recruitment and enrollment phase to the last evaluations, will last approximately 12 weeks.

   Participants will be enrolled as they accept and consent to have participated in the study. Once enrolled, the intervention will begin the following week, in order to reduce, as much as possible, the possibility of variation in the results of their initial measurements, between the previous evaluation period and the beginning of the intervention.
6. Intervention All participants in the intervention group will be assigned to one of two possible groups that will be developed in parallel, until completing the 8 weeks of intervention. The mindfulness intervention is based on the manual "Mindfulness Skills for Students" (provided and authorized for use by Dr Julieta Galante). This intervention consists of eight sessions of group mindfulness skills, carried out weekly by videoconference, each lasting 90 minutes. The sessions will be co-instructed by 3 facilitators. Two of them will direct the activities of the session and a third facilitator will have the role of technically helping to carry out the session, the monitoring of adverse events and eventual containment of the participants who need it.

Participants will receive the mindfulness application manual. In addition, they will be asked to practice daily at home, giving them access to an online platform via CANVAS with audiovisual material to guide their personal practice and they will also be asked to record their practice in the Home Practice Records that will be sent and completed. via CANVAS. The home practice questionnaires will ask what mindfulness skills were practiced and the number of minutes practiced. Participants will be asked to attend all eight sessions. Session attendance data will be collected and evaluated.

Mindfulness skills to be taught will include sitting meditation with mindfulness of breath, thoughts, emotions, or physical sensations; body scan meditation; standing meditation; and attention to routine daily activities. The didactic content will be presented and discussed in the group, with content focused on topics on how to define mindfulness and how it can help with stress and pain management, the difference between mindfulness and being on "automatic pilot", the stress, how our perceptions affect stress, the relationship between pain-suffering and distressing thoughts and emotions, the acceptance of pain and unwanted experiences, the use of mindfulness in daily life.

6.1. Control group Control group participants will enter a waiting list, and will cease to be in this condition once the study is completed (end of post-intervention evaluation). Then they will be offered to participate in the same intervention offered to the participants of the intervened group, with the same team of facilitators. During this stage there will only be an evaluation of potential adverse events during the sessions, and the same protocol mentioned for these purposes in the description of the intervention will be followed. There will be no evaluation of the symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students from the Universidad de los Andes, studying from 2nd to last year of undergraduate studies.
* Over 18 years.
* Able to read and speak Spanish.
* Scored on the PHQ-9 depression scale ≤ 14.
* Have participated in an informative meeting about the study and the implications of the intervention.
* Availability of time to participate in 1 weekly session of 90 minutes, for 8 consecutive weeks, and time to perform mindfulness exercises at home for at least 15 minutes a day, during the duration of the intervention.

Exclusion Criteria:

* With a PHQ-9 score greater than or equal to 15
* With active suicidality, defined as suicidal ideation, planning or attempt, or self-injurious behavior in the last 12 months.
* History of psychiatric treatment for a serious condition, understood as: psychotic pathology and / or substance abuse.
* History of hospital admission for psychiatric pathology, in the last 2 years.
* History of having participated in a previous Mindfulness-based course, such as: MBCT, MBSR, MMB, among others.
* History of severe trauma or sexual abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability and satisfaction | 1 week
  To determine the acceptability and satisfaction of the participants with the intervention using the Client Satisfaction Questionnaire (CSQ-8) of the intervention. The CSQ-8 is an instrument validated in English, and translated and validated into Spanish of 8 items that measures general satisfaction with health services received in different populations. The responses are of the Likert type with 4 options each. The questions are: How would you rate the services received? Did you receive the kind of service you required? To what extent has our program helped solve your problems? If a friend were in need of similar help, would you recommend our program? How satisfied are you with the amount of help you have received? Have the services you received helped you better deal with your problems? Overall, how satisfied are you with the services you have received? If you needed help again, would you return to our program? In addition, it has space to write down comments and suggestions.
Feasibility assessment | 12 weeks
  To determine the feasibility of study subject recruitment, participant retention, session attendance, and quantitative and qualitative data collection during an 8-week MBCT online program

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 12 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the 9 DSM-IV criteria from "0" (Never) to "3" (Almost every day). In Chile, it has validation for the detection of Chilean people aged 20 years and over, with a sensitivity of 92% and a specificity of 89%, compared to the Hamilton Depression scale. Furthermore, it has construct validity and predictive validity concurrent with the ICD-10 criteria for depression. It has 9 items. The interpretation is made by adding the total of the 9 questions as follows: 1-4 points, Minimal depression; 5-9, Medium depression; 10-14, Moderate depression; 15-19, moderately severe depression; 20-27, Severe depression.
Generalized Anxiety Disorder 7 (GAD-7) | 12 weeks
  The Generalized Anxiety Disorder 7 is an instrument developed from the PRIME-MD diagnostic instrument for common mental disorders. This consists of 7 questions. The score is calculated by assigning scores from 0 to 3, to the response categories from "Never" to "Almost every day." The total GAD-7 score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-off points for mild, moderate, and severe anxiety, respectively. It has been validated in Spanish, where a cut-off score of 10 showed adequate sensitivity (86.8%) and specificity (93.4%) values.
The alcohol, smoking and substance involvement screening test (ASSIST) | 12 weeks
  The ASSIST evaluates the use 10 substances: tobacco, alcohol, cannabis, cocaine, amphetamines, inhalants, sedatives, hallucinogens, opioids, and "other drugs". It is an instrument validated as an interview, in multiple languages; it has 8 questions covering frequency and associated problems for each substance. Although this instrument is only validated as a face-to-face interview, it will be adapted to a self-report due to its high acceptability in the literature and comprehensibility regarding the subject evaluated.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health v1.2 | 12 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS®) is an initiative of the National Institute of Health to develop measures that assess function and well-being in the domains of physical, mental and social health. It has been translated into multiple languages and multiculturally validated. This instrument assesses 5 areas: physical function, pain, fatigue, emotional stress and social health. 4 items are used to assess overall physical health, 3 of which use 5-category scales, and one item uses a scale of 1-10. 4 items are used to assess overall mental health, all using 5-category scales.
Five Facet Mindfulness Questionnaire (FFMQ) | 12 weeks
  The original questionnaire in English is a 39-item self-report that measures Mindfulness from five facets called Observation, Description, Acting with Consciousness, Absence of Judgment and Absence of Reactivity. Participants must answer each item on a Likert scale with a range from 1 (never or very rarely true) to 5 (very often or always true); The minimum score for the Questionnaire is 39 points and the maximum is 195 points. The instrument has adequate to good levels of reliability (Cronbach's alpha from .75 to .92). In Chile, the questionnaire was translated into Spanish and retranslated by bilingual psychologists, then it was applied in a pilot with high experience in the practice of meditation, with a validation in Chile.
Medical Outcome Study (MOS) Short Form (SF-36 v.2) | 12 weeks
  The SF-36 v.2 evaluates quality of life and general health status. It was developed by the Medical Outcome Study (MOS) and contains 36 items that are grouped into 8 health domains (Physical Function, Physical Role, Body Pain, General Health, Vitality, Social Function, Emotional Role, and Mental Health). The results of each of the dimensions are coded and transformed on a scale that ranges from 0 (the worst state of health) to 100 (the best state of health), and although the questionnaire is not designed to give a global index, it allows the calculation of two summary scores: Physical and Mental. This instrument has a validation in Chile.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete Olivares, MD, PhD, Principal Investigator — Universidad de Los Andes
Locations (1):
- Universidad de los Andes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
No share of individual participant data is planned because of restrictions provided by the Ethical Committee.

REFERENCES:
- [Background] Gili M, Castellvi P, Vives M, de la Torre-Luque A, Almenara J, Blasco MJ, Cebria AI, Gabilondo A, Perez-Ara MA, A MM, Lagares C, Pares-Badell O, Piqueras JA, Rodriguez-Jimenez T, Rodriguez-Marin J, Soto-Sanz V, Alonso J, Roca M. Mental disorders as risk factors for suicidal behavior in young people: A meta-analysis and systematic review of longitudinal studies. J Affect Disord. 2019 Feb 15;245:152-162. doi: 10.1016/j.jad.2018.10.115. Epub 2018 Oct 26. PMID 30390504
- [Background] Slavin SJ, Schindler DL, Chibnall JT. Medical student mental health 3.0: improving student wellness through curricular changes. Acad Med. 2014 Apr;89(4):573-7. doi: 10.1097/ACM.0000000000000166. PMID 24556765
- [Background] Hope V, Henderson M. Medical student depression, anxiety and distress outside North America: a systematic review. Med Educ. 2014 Oct;48(10):963-79. doi: 10.1111/medu.12512. PMID 25200017
- [Background] Hofmann SG, Gomez AF. Mindfulness-Based Interventions for Anxiety and Depression. Psychiatr Clin North Am. 2017 Dec;40(4):739-749. doi: 10.1016/j.psc.2017.08.008. Epub 2017 Sep 18. PMID 29080597
- [Background] Demarzo M, Montero-Marin J, Puebla-Guedea M, Navarro-Gil M, Herrera-Mercadal P, Moreno-Gonzalez S, Calvo-Carrion S, Bafaluy-Franch L, Garcia-Campayo J. Efficacy of 8- and 4-Session Mindfulness-Based Interventions in a Non-clinical Population: A Controlled Study. Front Psychol. 2017 Aug 8;8:1343. doi: 10.3389/fpsyg.2017.01343. eCollection 2017. PMID 28848465
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Background] Blanck P, Perleth S, Heidenreich T, Kroger P, Ditzen B, Bents H, Mander J. Effects of mindfulness exercises as stand-alone intervention on symptoms of anxiety and depression: Systematic review and meta-analysis. Behav Res Ther. 2018 Mar;102:25-35. doi: 10.1016/j.brat.2017.12.002. Epub 2017 Dec 20. PMID 29291584
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Cebolla A, Demarzo M, Martins P, Soler J, Garcia-Campayo J. Unwanted effects: Is there a negative side of meditation? A multicentre survey. PLoS One. 2017 Sep 5;12(9):e0183137. doi: 10.1371/journal.pone.0183137. eCollection 2017. PMID 28873417
- [Background] Blatch-Jones AJ, Pek W, Kirkpatrick E, Ashton-Key M. Role of feasibility and pilot studies in randomised controlled trials: a cross-sectional study. BMJ Open. 2018 Sep 25;8(9):e022233. doi: 10.1136/bmjopen-2018-022233. PMID 30257847